CLINICAL TRIAL: NCT01516060
Title: The Neurocognitive Sub Study of Encore1:A Randomised, Double-Blind, Placebo-Controlled, Clinical Trial to Compare the Safety and Efficacy of Reduced Dose Efavirenz (EFV) With Standard Dose EFV Plus 2N(t)RTI in Antiretroviral-naïve HIV-Infected Individuals Over 96 Weeks A Randomised, Double-blind, Placebo-controlled, Clinical Trial to Compare the Safety and Efficacy of Reduced Dose Efavirenz (EFV) With Standard Dose EFV Plus Two Nucleotide Reverse Transcriptase Inhibitors (N(t)RTI) in Antiretroviral-naïve HIV-infected Individuals Over 96 Weeks
Brief Title: The Neurocognitive Sub-study of Encore1
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Kirby Institute (Other Government)
Collaborators: The HIV Netherlands Australia Thailand Research Collaboration (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Screening
Other Study IDs: Encore1-NC
Record Dates: First submitted 2012-01-19; First posted 2012-01-24 (Estimated); Last update posted 2013-09-19 (Estimated); Status verified 2013-09

CONDITIONS: HIV
MeSH Terms: interventions — efavirenz

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Reduced dose Efavirenz arm (Experimental): Patient's on main study that was randomised to receive TDF (300mg qd)/FTC (200mg qd) + EFV (400mg qd; 2 x 200mg + 1 x 200mg placebo qd).
  Interventions: Drug: Efavirenz
- Normal Efavirenz dose arm (Active Comparator): Patient's on main study randomised to receive tenofovir (TDF) (300mg qd)/emtricitabine (FTC) (200mg qd) + EFV (600mg qd; 3 x 200mg qd)
  Interventions: Drug: Efavirenz

INTERVENTIONS:
Drug: Efavirenz — 400mg qd; 2 x 200mg
  Arms: Reduced dose Efavirenz arm
Drug: Efavirenz — 600mg qd; 3 x 200mg qd
  Arms: Normal Efavirenz dose arm

SUMMARY:
The purpose is to investigate whether HIV and HIV medication can affect certain areas of brain function. This study will look at possible changes in brain function including memory, concentration and thought processes to see if there are any differences between the two doses of efavirenz used in the Encore1 study and also the level of efavirenz in the blood

ELIGIBILITY:
Inclusion Criteria:

* All subjects entering into the main study protocol at participating centres will be eligible to enter this sub-study.

Exclusion Criteria:

* Existing neurological brain disease
* Recent (<6months ) head injury
* Current major depression or psychosis
* Current alcohol abuse
* Intended use of recreational drugs during study period
* Uncontrolled medical conditions deemed to potentially interfere with cognitive function (e.g. uncontrolled diabetes, pyrexial illness, uraemia etc)

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 71 (Actual)
Dates: Start 2012-01; Primary Completion 2013-03 (Actual); Study Completion 2013-03 (Actual)

PRIMARY OUTCOMES:
The primary endpoint is the comparison between of neurocognitive function in patients initiating sdEFV and 400EFV | 48 weeks

SECONDARY OUTCOMES:
The association between week 4 plasma EFV levels and change from baseline neurocognitive function to week 4 and 24. | Week 24
To assess dynamic changes in neurocognitive function over the total duration of follow-up. | 96 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Rebekah Puls, Principal Investigator — Kirby Institute
Locations (1):
- HIVNAT Research Collaboration, Bangkok, Thailand